CLINICAL TRIAL: NCT00483119
Title: Phase 2 Randomized Trial of IVIg With or Without Cyclophosphamide in Pemphigus
Brief Title: Randomized Trial of IVIg With or Without Cyclophosphamide in Pemphigus
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to the death of the PI.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3343
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Results first posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-01

CONDITIONS: Pemphigus Vulgaris
Keywords: pemphigus vulgaris; IVIg; cyclophosphamide; treatment; pemphigus antibodies
MeSH Terms: conditions — Pemphigus | interventions — Immunoglobulins, Intravenous; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Active Comparator): IVIg alone (intravenous immunoglobulin)
  Interventions: Drug: intravenous immunoglobulin
- Group B (Experimental): IVIg with cyclophosphamide
  Interventions: Drug: intravenous immunoglobulin; Drug: cyclophosphamide

INTERVENTIONS:
Drug: intravenous immunoglobulin — Gamunex 10% 500/mg/kg/day x four days per cycle total of four cycles
  Other Names: IVIg; Gamunex
Drug: cyclophosphamide — cyclophosphamide dose of 2mg/kg/day divided into three-times daily oral administration
  Other Names: CP
  Arms: Group B

SUMMARY:
The purpose of this study is to compare two standard treatments for pemphigus to determine which more effectively improves the clinical manifestations of the disease and decreases serum level of the autoantibodies which cause the disease.

DETAILED DESCRIPTION:
Pemphigus is a serious and life-threatening autoimmune disease characterized by blisters and erosions that occur on the skin and oral mucosa. It is caused by autoantibodies that attack desmoglein 1 and 3, adhesion molecules that are present on the surface of the cells (keratinocytes) that make up the superficial layer of the skin. As a result these cells stop sticking together, and come apart resulting in the formation of blisters on the skin.

Pemphigus is usually treated with systemic corticosteroids often given together with immunosuppressive drugs such as Cytoxan (cyclophosphamide), Imuran (azathioprine), methotrexate, CellCept (mycophenolate mofetil) and others. However, the prolonged and high doses of systemic steroids and other immunosuppressive agents used to treat the disease are associated with significant toxicity.

A new treatment which is now being used to treat pemphigus patients that are unresponsive, or that have developed complications to conventional treatment is IVIg (intravenous immunoglobulin). IVIg consists of one of the protein fractions present in blood. It is the fraction that contains antibodies and is called immunoglobulin (Ig). It is purified from blood that has been collected from thousands of donors and treated to remove potential infectious agents. It is administered intravenously (IV) over several hours, several days in succession. The cycles are usually repeated every 2 to 4 weeks until the disease is controlled.

IVIg treatment is currently given in either of two ways, either by itself or with an immunosuppressive drug such as cyclophosphamide or azathioprine. It is unknown which of these two procedures is better. This trial is being conducted to determine which treatment is more effective.

The trial is being conducted in patients with pemphigus that are not responding to, or have developed complications from, standard treatment. All patients will be treated with IVIg administered using a standard protocol. The IVIg will be given daily for 4 days, and this cycle will be repeated every other week for a total of 4 cycles. In addition, half of the patients will be selected by chance to also be treated with cyclophosphamide, an immunosuppressive drug often used to treat other autoimmune diseases including pemphigus. The cyclophosphamide is a pill that is taken 3 times a day. A total of 12 patients will be treated in each arm of the trial. The trial is being conducted by Dr. Jean-Claude Bystryn at the New York University Medical Center.

The extent and activity of the disease, as well as the blood levels of pemphigus antibodies, will be measured at baseline prior to entry into the trial and periodically during the trial.

The goal of the study is to determine whether there is a difference between the two treatments in the rate at which: 1) the activity and extent of the disease improves, 2) the dose of corticosteroids required to treat the disease can be reduced, and 3) the blood level of pemphigus antibodies decrease.

This trial will test this hypothesis by examining whether IVIg treatment given with cyclophosphamide results in a more rapid decline in circulating pemphigus antibodies than when given alone.

ELIGIBILITY:
Inclusion Criteria:

* Lesions consistent with pemphigus foliaceus or vulgaris
* Diagnosis confirmed by histology and IIF ≥ 40 within past month
* On ≥20mg/day of prednisone per day for two weeks or ≥ 80mg/day for one week
* Women of childbearing potential negative HCG obtained two weeks prior to first IVIg
* Agrees to two acceptable forms of contraception* if randomized to cyclophosphamide group:
* IUD (except progesterone T), Combination oral contraceptives, transdermal patch, vaginal ring, hormonal injectables or implantables, male latex condom, diaphragm, cervical cap, or vaginal sponge (contains spermicide)
* Normal organ function confirmed by CBC, UA, LFTs and Ig levels within defined inclusion criteria
* Responds yes to at least one of the criteria below:
* Persistence of clinical manifestations of disease despite steroid treatment
* Flare in disease activity after an attempt at steroid tapering
* Failure of established lesions to heal
* Rapidly progressive disease.
* Conventional therapy is relatively contraindicated i.e. side effects, co-morbid conditions
* systemic infections, peptic ulcers, osteoporosis, hypertension, cataracts or others

Exclusion Criteria:

* Use of IVIg within past 3 weeks or the use of a cytotoxic drug within the past 2 weeks
* Participating in another clinical trial at the time of screening and enrollment
* Medical condition that precludes use of IVIg or cyclophosphamide (i.e. pregnancy breastfeeding, underlying chronic infection, concurrent opportunistic infection, sepsis or volume depletion
* Renal insufficiency ( GFR <90, proteinuria (>1+, x 2), creatinine >1.8 or increased WBC or RBCs which cannot be explained by cystitis.)
* Known hypersensitivity to study drugs, IVIg or cyclophosphamide

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Bystryn, M.D., Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- NYU Medical Center, New York, New York, United States

REFERENCES:
- [Background] Green MG, Bystryn JC. Effect of intravenous immunoglobulin therapy on serum levels of IgG1 and IgG4 antidesmoglein 1 and antidesmoglein 3 antibodies in pemphigus vulgaris. Arch Dermatol. 2008 Dec;144(12):1621-4. doi: 10.1001/archdermatol.2008.503. PMID 19075146
- [Background] Czernik A, Bystryn JC. Kinetics of response to conventional treatment in patients with pemphigus vulgaris. Arch Dermatol. 2008 May;144(5):682-3. doi: 10.1001/archderm.144.5.682. No abstract available. PMID 18490602
- [Background] Czernik A, Beutner EH, Bystryn JC. Intravenous immunoglobulin selectively decreases circulating autoantibodies in pemphigus. J Am Acad Dermatol. 2008 May;58(5):796-801. doi: 10.1016/j.jaad.2008.01.007. PMID 18423257
- [Background] Czernik A, Bystryn JC. Improvement of intravenous immunoglobulin therapy for bullous pemphigoid by adding immunosuppressive agents: marked improvement in depletion of circulating autoantibodies. Arch Dermatol. 2008 May;144(5):658-61. doi: 10.1001/archderm.144.5.658. PMID 18490594

RESULTS

PARTICIPANT FLOW:
Groups:
- IVIg Alone: IVIg alone
  intravenous immunoglobulin: Gamunex 10% 500/mg/kg/day x four days per cycle total of four cycles
- IVIg With Cyclophosphamide: IVIg with cyclophosphamide
  cyclophosphamide: cyclophosphamide dose of 2mg/kg/day divided into three-times daily oral administration
Period: Overall Study
Arm/Group | IVIg Alone | IVIg With Cyclophosphamide
Started | 5 | 4
Completed | 4 | 3
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: This number is based only on the number of patients who passed screening and then were enrolled. Please note that this study was not evaluable due to the untimely death of the study Principal Investigator as noted previously.
Groups:
- Group A: IVIg alone
  intravenous immunoglobulin: Gamunex 10% 500/mg/kg/day x four days per cycle total of four cycles
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 4 | 3 | 7
Age, Continuous [Mean (Full Range); unit: years] | 61.2 [45 to 68] | 56.25 [47 to 66] | 59 [45 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Clinical Outcome: Extent and Severity of Disease
Time Frame: 6 - 10 weeks after initiation of therapy
Population: Sadly, the trial PI, Dr. Jean-Claude Bystryn, died on August 19, 2010. As a result the study could not be completed and an analysis of the data collected was not performed.
Arm/Group | IVIg Alone | IVIg With Cyclophosphamide
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Serum Levels of Pemphigus Antibodies
Time Frame: 6-10 weeks after initiation of therapy
Population: as for outcome 1
Arm/Group | IVIg Alone | IVIg With Cyclophosphamide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Toxicity of Treatment: Measured in Renal Toxicity, Myelosuppression or Hepatic Toxicity
Time Frame: Throughout course of study
Population: as for outcome 1
Arm/Group | IVIg Alone | IVIg With Cyclophosphamide
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Ability to be Weaned Off Steroids
Time Frame: Measured 6 and 10 weeks after initiation of IVIg treatment
Population: as for outcome 1
Arm/Group | IVIg Alone | IVIg With Cyclophosphamide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=5) | Group B (N=4)
Atrial Fibrillation not considered related to treatment (Cardiac disorders) | 0 (0) | 1 (1) — event occurred 5 days post infusion
Elevated blood pressure; blurred vision, nausea and tearing (Cardiac disorders) | 1 (1) | 0 — Day 3 of IVIG infusion cycle 3; At the infusion suite his blood pressure was 160/106 mmHg and the headache was still persistent. IVIG was not infused. Patient was sent to NYULMC ER for evaluation. Brain CT was normal. Patient withdrawn from study.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=5) | Group B (N=4)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Chest Tightness (Cardiac disorders) | 1 (1) | 0 (0) — Intermittant following infusion for 2 hours
Increased Creatine Levels (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 4 (4) | 0 (0)
Mild Muscle Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Elevated Urine Protein Levels (Renal and urinary disorders) | 2 (2) | 0 (0) — Creatine levels remained normal throughout event.
Localized minor inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — At infusion site.
Pulmanary Adema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oral Candida Infection (Infections and infestations) | 0 (0) | 1 (1)
leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1) | 1 (1)
Mild Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mild skin infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Penile Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Vasovega (Nervous system disorders) | 1 (1) | 0 (0)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Food Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Sadly, the trial PI, Dr. Jean-Claude Bystryn, died on August 19, 2010. As a result the study could not be completed and an analysis of the data collected was not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No